CLINICAL TRIAL: NCT01952509
Title: Multinational, Multicenter, Non Interventional Study, in Patients With Rheumatoid Arthritis (RA) Treated With Tocilizumab.
Brief Title: A Non-Interventional Study of RoActemra/Actemra (Tocilizumab) Treatment in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28747
Record Dates: First submitted 2013-09-10; First posted 2013-09-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, observational study will evaluate the use and efficacy of RoActemra/Actemra (tocilizumab) in routine clinical practice in patients with moderate to severe rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment in accordance with the local label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patients in whom the treating physician has made the decision to commence RoActemra/Actemra treatment (in accordance with the local label); this can include patients who have received RoActemra/Actemra treatment within 8 weeks prior to the enrolment visit

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Patients who have received treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* Patients with a history of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe rheumatoid arthritis initiating treatment with RoActemra/Actemra in accordance with the local label
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on RoActemra/Actemra at 6 months after treatment initiation | approximately 2 years

SECONDARY OUTCOMES:
Rates of dose modifications/interruptions | approximately 2 years
Clinical/demographic patient characteristics at initiation of RoActemra/Actemra treatment | approximately 2 years
Proportion of patients on RoActemra/Actemra monotherapy at study entry and at Month 6 | approximately 2 years
Efficacy: Response according to total joint count evaluation by DAS28/EULAR/SDAI/CDAI/ACR | approximately 2 years
Safety: Incidence of adverse events | approximately 2 years
Health Assessment Questionnaire Disability Index | approximately 2 years
Visual Analogue Scale - Fatigue | approximately 2 years
Visual Analogue Scale - severity of pain | approximately 2 years
Visual Analogue Scale - morning stiffness | aproximately 2 years
Patient Global Assessment of disease activity | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Costa Rica (2):
  - Cartago
  - San José
- Santo Domingo, Dominican Republic
- Guatemala City, Guatemala
- Panama City, Panama